CLINICAL TRIAL: NCT06151327
Title: Explore the Relationship Between Implementation of Alternating Pressure Air Mattress and Pressure Injury Prevalence
Brief Title: Alternating Pressure Air Mattress and Pressure Injury Prevalence
Acronym: APAM
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202309095RINA
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pressure Injury; Alternating Pressure Air Mattress; Implementation
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
explore the correlation of accurate implementation of APAM and pressure injury prevalence

ELIGIBILITY:
Inclusion Criteria:

patients with pressure injury

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients in hospital with pressure injury
Sampling Method: Non-Probability Sample
Enrollment: 50419 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
proportion of full thickness pressure injury | 2020/1 ~2023/8
  total number of full thickness pressure injuries devided by total number of pressure injuries

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsiu Chang, Principal Investigator — National Taiwan University Hospital Yunlin brach
Locations (1):
- National Taiwan Universiyt Hospital Yunlin Branch, Douliu, Yunlin, Taiwan